CLINICAL TRIAL: NCT03422809
Title: Cyclic Variation in Micronutrient Concentrations and Plasma Volume in Reproductive-Age Women
Brief Title: Cyclic Variation in Micronutrient Concentrations and Plasma Volume
Status: Completed | Type: Observational
Sponsor: Alison Gernand (Other)
Collaborators: Penn State University (Other)
Responsible Party: Sponsor-Investigator, Alison Gernand, Assistant Professor of Nutritional Sciences, Penn State University
Organization: Penn State University (Other)
Other Study IDs: STUDY00008383
Record Dates: First submitted 2018-01-16; First posted 2018-02-06 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Plasma Volume; Micronutrients; Menstrual Cycle
Keywords: Plasma volume, micronutrient, estrogen, progesterone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, serum and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall goal of this study is to examine the influence of the menstrual cycle on micronutrient concentrations and plasma volume in healthy, reproductive-age women with regular cycles. The investigators aim to quantify changes in micronutrient biomarker concentrations (zinc, copper, iron, and vitamin A) and plasma volume across the menstrual cycle in healthy women.

DETAILED DESCRIPTION:
This is a longitudinal prospective study wherein all subjects will be examined at three time points within a single menstrual cycle: the early follicular phase (~day 2), periovulation (~day 12), and the luteal phase (~day 21)-based on an approximate 28-day cycle length. The actual days of visits will be adjusted for the length of the woman's menstrual cycle. At least 35 non-pregnant women ages 18 to 44 years will be recruited as a convenience sample of eligible women in the State College area and surrounding towns within Centre County, Pennsylvania, USA. If a woman responds to the recruitment, she will be asked a set of pre-screening questions to determine eligibility. If a woman is thought to be eligible, she will complete a verbal consent for the screening (and the actual screening will occur at the first visit). Then she will be invited to the Clinical Research Center (CRC), a service unit in Penn State's Clinical and Translational Science Institute, for full screening and participation. Before scheduling the visit, the woman will be asked for the expected date of the first day of her next menstrual period. The woman will then be tentatively scheduled for her first visit at the CRC approximately 1 day after this date (avoiding weekend days).

As part of the preparation for study visits, the woman will be asked to fast the night before her visit. Women will also be asked to avoid alcohol intake for 12 hours preceding their scheduled visits to the CRC, and to drink plenty of water. On the morning of the visit, the woman will arrive at the CRC, go through complete screening (including height, weight, blood pressure, and pregnancy test). If eligible for the main study, the woman will then go through the consent process for the main study. If the woman gives consent to participate, the investigators will then proceed with study measurements (including a questionnaire and body composition measurement).

Following these measurements, the study nurse or doctor will insert an IV into the vein of one arm and an initial baseline blood draw will be taken (~15-20 ml, in several tubes). This blood will be used for biomarker assessment (hemoglobin, hematocrit, vitamins, minerals, etc) and as a blank sample before the dye injection. Next, indocyanine green (ICG) will be used to measure plasma volume. A solution will be prepared using 25 mg of ICG lyophilized powder dissolved in 10 ml of sterile water. The investigators will draw enough solution to inject 0.25 mg/kg body weight into a syringe. The syringe will be weighed to measure the exact amount. Then the solution will be injected via the IV and flushed with saline. After 2 minutes, five ~3 ml blood samples will be drawn at intervals of 45 seconds over the next 3 minutes. Expected total volume of blood drawn at the visit will be <35 mL.

At the end of this first visit the participant will be given a home-based fertility monitor to take home to track her cycle. She will be instructed on how to use the monitor at home but the research team will maintain contact with her on a regular basis to ensure that she is using the monitor correctly. She will conduct a daily urine test with the monitor, which uses urine hormone concentrations to track the stage of the menstrual cycle for the participants by displaying low, high, or peak fertility. The second and third visits will be scheduled using an algorithm that takes into consideration the woman's menstrual cycle length and results from a home-based urine fertility monitor.

At the third visit, the participant will return the monitor to the CRC and the urine test results, which are stored in the monitor, will be retrieved. At the end of the third visit her study participation is complete but the investigators will keep in contact with her to record the first date of her next cycle (to calculate actual cycle length).

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 to 44 years of age
* General good health (does not have a known, ongoing health condition/medical issue that requires regular monitoring by a doctor or regular visits to the hospital)
* BMI 18.5-24.9 kg/m2
* Regular menstrual cycle (26-35 days)
* Non-smoker
* Non-pregnant
* If pregnant before, ≥12 months since last pregnancy

Exclusion Criteria:

* Known allergy to shellfish or iodine
* Blood pressure on the day of measurements is low or high (systolic blood pressure (SBP) <90 or ≥130 mmHg and/or diastolic blood pressure (DBP) <60 or ≥80 mmHg)
* Currently has low or high blood pressure (SBP <90 or ≥130 mmHg and/or DBP <60 or ≥80 mmHg), self-reported
* Current hypertension or previous hypertensive disorder in pregnancy (gestational hypertension or preeclampsia)
* Taking regular medication(s) (physician's prescribed medications for a health condition)
* Currently trying to conceive
* Currently breastfeeding
* Currently using hormonal birth control or used within last 3 months
* Used depot medroxyprogesterone acetate (DMPA) in the past 12 months
* Diagnosis of polycystic ovary syndrome

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participant eligibility is based on biological description of gender identity.
Study Population: Eligible women in the State College area and surrounding towns within Centre County, Pennsylvania, United States.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Change in serum zinc concentration across the menstrual cycle | ~3 weeks (~day 2 to day ~21 of a 28 day menstrual cycle)
  Difference in mean serum zinc concentrations measured at three time points (day ~2, day~12 and day~21) within a single menstrual cycle will be examined.
Change in serum copper concentration across the menstrual cycle | ~3 weeks (~day 2 to day ~21 of a 28 day menstrual cycle)
  Difference in mean serum copper concentrations measured at three time points (day ~2, day~12 and day~21) within a single menstrual cycle will be examined.
Change in serum retinol concentration across the menstrual cycle | ~3 weeks (~day 2 to day ~21 of a 28 day menstrual cycle)
  Difference in mean serum retinol concentrations measured at three time points (day ~2, day~12 and day~21) within a single menstrual cycle will be examined.
Change in plasma volume across the menstrual cycle | ~3 weeks (~day 2 to day ~21 of a 28 day menstrual cycle)
  Difference in mean plasma volume measured at three time points (day ~2, day~12 and day~21) within a single menstrual cycle will be examined.

SECONDARY OUTCOMES:
Change in serum ferritin concentration across the menstrual cycle | ~3 weeks (~day 2 to day ~21 of a 28 day menstrual cycle)
  Difference in mean serum ferritin concentrations measured at three time points (day ~2, day~12 and day~21) within a single menstrual cycle will be examined.
Change in hemoglobin concentration across the menstrual cycle | ~3 weeks (~day 2 to day ~21 of a 28 day menstrual cycle)
  Difference in mean hemoglobin concentrations measured at three time points (day ~2, day~12 and day~21) within a single menstrual cycle will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Gernand, PhD, Principal Investigator — The Pennsylvania State University
Locations (1):
- The Pennsylvania State University, State College, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No